CLINICAL TRIAL: NCT02451254
Title: Coagulation Activity and Thrombogenesis in Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Tel-Aviv Sourasky Medical Center, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-15-EC-0142-15-CTIL
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atrial Fibrillation (Experimental): Atrial Fibrillation patients electively admitted for circumferential ablation of the pulmonary veins.
  Interventions: Procedure: circumferential ablation
- control (Active Comparator): patients electively admitted for SVT ablation
  Interventions: Device: SVT ablation

INTERVENTIONS:
Procedure: circumferential ablation — circumferential ablation of the pulmonary veins
  Arms: Atrial Fibrillation
Device: SVT ablation — SVT ablation
  Arms: control

SUMMARY:
Atrial fibrillation confers up to 5-fold increased risk of stroke in the absence of valvular heart disease. Although epidemiological studies have linked various clinical and echocardiographic risk factors to stroke, the exact mechanism of increased risk of stroke in AF remains poorly understood. Previous reports have suggested that loss of effective atrial contraction because of AF is associated with thrombogenesis. Microthrombi are most likely to form in the left atrial appendage. In contrast, intravascular thrombotic events in patients without AF are generally associated with abnormalities of vascular endothelial function and/or the coagulation system. On the assumption that more than 90% of all cardiac thrombi in patients with AF form in the LA appendage, and the fact that thrombi have been identified in 15-20% of patients with AF who have clinical risk factors for ischemic stroke, it has been deemed to be "our most lethal attachment". Administration of anticoagulant therapy is generally thought to be necessary as a preventive measure for patients at high risk of thromboembolism, but data indicating inadequate implementation of this highly effective therapy]. Several studies have found regional differences in platelet activation and hypercoagulability in the LA compared with systemic circulation in patients with valvular and nonvalvular AF, suggesting local contributing factors. Animal studies have demonstrated increased platelet activation and endothelial dysfunction with acute AF. The ability of antiplatelet agents to reduce the risk of cardioembolic events in AF suggests that platelets may contribute to the pathophysiology. Platelet activation occurs with AF and rapid atrial pacing, providing a possible mechanistic link. Other biomarkers that have proposed to improve the prediction of thromboembolotic events in this patient population include von Willebrand factor and D-dimer and cerebral imaging. A comprehensive understanding of the pathophysiological sequence leading to thrombus formation in the LAA of patients with AF could be helpful to characterize those at high risk for thromboembolic events, and subsequently to optimize the management of high risk patients.

DETAILED DESCRIPTION:
Aim: To compare biomarkers and mediators associated with arterial and venous thrombosis from blood sampling from the LA, RA, and systemic circulation in patients with AF.

Methods and population: A prospective trial of patients who undergo circumferential ablation of the pulmonary veins. For the clinical procedure, a conventional transeptal puncture is performed. In the beginning of the procedure, following transeptal puncture, and before intravenous administration of unfractionated heparin (bolus of 50-100 IU/kg), blood samples will simultaneously be collected from the peripheral femoral venous sheath, arterial line, right atrial sheath, and LA sheath. Samples from the RA and LA will be collected with the sheath positioned in the midchamber and close to the appendages. Each Patient will provide up to 40ml of blood for the following blood tests: (1) Blood count. (2) Fibrinogen (3) Factor VIII (4) D-dimer (5) P-selectin (6) von Willebrand factor (7) TEG - Thromboelastography Serum and plasma samples will be stored for future tests.

ELIGIBILITY:
Inclusion Criteria:

1. AF patients from cardiology department in our institution electively admitted for circumferential ablation of the pulmonary veins.
2. Control - patients from cardiology department in our institution electively admitted for SVT ablation.

Exclusion Criteria:

1.Intra- and extra-cardiac shunts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Thrombotic biomarkers in AF patients | 12 months
  comparison of blood sampling from the LA, RA, and systemic circulation in AF patients

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Chorin, MD, Principal Investigator — Tel Aviv Medical Center
Locations (2):
- Israel (2):
  - Tel Aviv medical center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No